CLINICAL TRIAL: NCT02739256
Title: Normal Voiding Function After Surgical Repair of Pelvic Organ Prolapse: A Randomized Trial Comparing Day of Surgery Retrograde Void Trials to Standard Postoperative Day One Retrograde Void Trials
Brief Title: Early Versus Late Voiding Trials After Prolapse Repair
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Institutional implementation of a same day discharge pathway
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Charelle Carter-Brooks, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PRO15100653
Record Dates: First submitted 2016-03-10; First posted 2016-04-15 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Urinary Retention; Pelvic Organ Prolapse
Keywords: voiding trial; pelvic organ prolapse; post-operative catheterization
MeSH Terms: conditions — Urinary Retention; Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- voiding trial 4 hours post-op (Experimental)
  Interventions: Procedure: Retrograde voiding trial
- voiding trial post-op day 1 (Active Comparator)
  Interventions: Procedure: Retrograde voiding trial

INTERVENTIONS:
Procedure: Retrograde voiding trial — A bladder test is performed after surgery for prolapse to make sure the patient can empty their bladder prior to discharge from the hospital. The test consists of filling the bladder with 300 mL of water and removing the catheter. Then the patient voids.
  Other Names: Bladder Test

SUMMARY:
The primary aim of this study is to determine if normal bladder function (the ability to empty the bladder during spontaneous urination) after surgical repair of pelvic organ prolapse returns faster in patients who have a retrograde voiding trial the day of surgery versus patients who have a retrograde voiding trial on postoperative day one. Half of participants will have a voiding trial 4 hours after surgery, while the other half will have the voiding trial postoperative day one.

DETAILED DESCRIPTION:
Overnight indwelling catheterization is a prevalent practice after surgical repair of pelvic organ prolapse. A voiding trial is performed postoperative day one to determine if urinary retention or abnormal bladder function exists. A significant number of patients ranging from 26-47% will require continued catheterization post-op for urinary retention in order to avoid injuries associated with over distention of the bladder and ureteral reflux.

This study aims to explore a strategy to reduce the length of catheterization post-operatively by testing the bladder at a closer interval to surgery. An earlier voiding trial may improve patient perioperative satisfaction and decrease catheter associated urinary tract infections. Additional benefits that may also be seen are earlier first ambulation and quicker achievement of post-op discharge milestones (pain control, ambulation with symptoms, oral intake tolerance and completion of a voiding trial). To date, few studies have attempted a day of surgery voiding trial in patients being admitted for repair of pelvic organ prolapse that requires an overnight admission.

ELIGIBILITY:
Inclusion Criteria:

* surgical management of pelvic organ prolapse requiring an overnight hospital admission

Exclusion Criteria:

* same day surgery
* non-ambulatory (allowed to use an assistive device)
* inability to provide informed consent, age < 21 years
* pregnancy or desire for future pregnancy
* systematic disease known to affect bladder function (Parkinson's disease, Multiple Sclerosis, Spina Bifida, spinal cord injury or trauma and neurogenic bladder)
* known preoperative urinary retention (defined as a post-void residual > 100mL)
* an untreated urinary tract infection at the time of surgery
* treatment at the time of surgery for urinary tract infection
* symptoms of urinary tract infection on the day of surgery

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-02; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
time to return of normal bladder function | 5 days

SECONDARY OUTCOMES:
time to first ambulation | 24 hours
anxiety level | 24 hours
  The State-Trait Anxiety Index anxiety inventory will be administered pre-operatively and at 4 different time point post-operatively to assess the patient's level of anxiety related to the catheter
pain level | 24 hours
  A pain scale will be administered pre-operatively and at 4 different time point post-operatively to assess the patient's level of anxiety related to the catheter
patient preference in the timing of the voiding trial | 24 hours
  a brief survey will be given 4 times during the hospital admission assess this
catheter associated urinary tract infections | 6 weeks
  medical records will be reviewed after discharge from the hospital for positive urine cultures

CONTACTS AND LOCATIONS:
Overall Officials: Charelle Carter-Brooks, MD, Principal Investigator — Urogynecology Fellow
Locations (1):
- Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oliphant SS, Lowder JL, Ghetti C, Zyczynski HM. Effect of a preoperative self-catheterization video on anxiety: a randomized controlled trial. Int Urogynecol J. 2013 Mar;24(3):419-24. doi: 10.1007/s00192-012-1868-y. Epub 2012 Jul 3. PMID 22752014
- [Result] Geller EJ, Hankins KJ, Parnell BA, Robinson BL, Dunivan GC. Diagnostic accuracy of retrograde and spontaneous voiding trials for postoperative voiding dysfunction: a randomized controlled trial. Obstet Gynecol. 2011 Sep;118(3):637-642. doi: 10.1097/AOG.0b013e318229e8dd. PMID 21860294
- [Result] Turner LC, Kantartzis K, Shepherd JP. Predictors of postoperative acute urinary retention in women undergoing minimally invasive sacral colpopexy. Female Pelvic Med Reconstr Surg. 2015 Jan-Feb;21(1):39-42. doi: 10.1097/SPV.0000000000000110. PMID 25185611
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246